CLINICAL TRIAL: NCT01720329
Title: A Randomized Controlled Trial of Probiotics to Prevent Influenza and Other Respiratory Infections in Residents of Long-term Care Facilities: A Pilot Study
Brief Title: Use of Probiotics to Prevent Influenza
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PPI-2012
Record Dates: First submitted 2012-10-15; First posted 2012-11-02 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Active Comparator): Participants randomized to probiotics will receive 2 capsules supplemented with 10 billion cfu of Lactobacillus rhamnosus GG on a daily basis for six months
  Interventions: Dietary Supplement: Probiotics
- Probiotic placebo (Placebo Comparator): Participants randomized to placebo will receive 2 capsules of matching placebo on a daily basis for six months
  Interventions: Other: probiotic placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Active comparator Arm. XXmls of XXX supplemented with XX of L. rhamnosus GG on a daily basis for six months
  Arms: Probiotics
Other: probiotic placebo — Placebo comparator arm -Participants randomized to placebo will receive XXmls of XXX G on a daily basis for 6 months.
  Arms: Probiotic placebo

SUMMARY:
The goal of this study is to assess the feasibility of randomizing residents of long-term care facilities to either probiotics or placebo to assess whether probiotics can reduce influenza and other viral laboratory confirmed respiratory infection.

DETAILED DESCRIPTION:
The goal of this study is to assess the feasibility of randomizing residents of long-term care facilities to either probiotics or placebo to assess whether probiotics can reduce influenza and other viral laboratory confirmed respiratory infection. The investigators will determine whether it is feasible to enroll residents and randomize them to a daily course of probiotics or placebo and monitor for influenza and other respiratory tract infections. In addition, the investigators will asses the feasibility of obtaining a nasal specimen for evaluation of the upper respiratory microbiome, measure antimicrobials, and deterioration in functional status. All aspects of the proposed trial will be assessed, including enrollment, randomization, respiratory infection surveillance, methods for outcome assessment, and event rates. The investigators will test the use of our data collection forms and data management strategy and will generate date to derive an appropriate sample size.

ELIGIBILITY:
Inclusion Criteria:

* nursing home residents, 65 years of age or older, in the Hamilton ON area

Exclusion Criteria:

* residents who are immunosuppressed (steroids or other immunosuppressives), have a hematologic malignancy, structural heart disease, gastroesophageal or intestinal injury and those are at increased risk of an endovascular infection will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2013-07; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
laboratory-confirmed influenza or other respiratory viral infection in participants in intervention arm of study | Participants will be assessed twice weekly for symptoms for 6 months. This will begin after they have been randomized to probiotics or placebo arms of the study
  this will be confirmed on the basis of reverse transcriptase Polymerase Chain Reaction(PCR)

SECONDARY OUTCOMES:
influenza like illness | Participants will be assessed twice weekly for 6 months after they have been randomized into probiotics or placebo
  influenza-like illness will be defined by the presence of fever, sore throat, and cough and will measure symptom severity
antimicrobial prescriptions | To be reviewed at the twice weekly assessments for 6 months following randomization
  courses of antimicrobials (name, does and duration) will be recorded by research nurse using information on the medication container or by contacting the prescribing physician if necessary. We will measure antibiotic associated diarrhea which we define as ≥ 3 liquid stools/d for at least two day.
physician visits for respiratory illness | The participant's MD patient record will be reviewed for visits during the 12 months following randomization
  information will be obtained from the attending physician
hospitalizations for lower respiratory infection or pneumonia | Patient will be asked during the twice weekly assessments about any hospitalizations, as well as consulting their MD, during the 6 months following randomization
  cause of hospitalizations will be assessed by the research nurse through interviews with the participants and reviews of hospital medical records. Deaths will be recorded using medical records

CONTACTS AND LOCATIONS:
Overall Officials: Mark Loeb, MD, Principal Investigator — McMaster University, Hamilton, ON, Canada
Locations (13):
- Canada (13):
  - The Clarion, Hamilton, Ontario
  - Pine Villa, Hamilton, Ontario
  - Arbour Creek, Hamilton, Ontario
  - Parkview Nursing centre, Hamilton, Ontario
  - Dundurn Place, Hamilton, Ontario
  - Shalom Village, Hamilton, Ontario
  - The Wellington, Hamilton, Ontario
  - Idlewyld Manor, Hamilton, Ontario
  - Regina Gardens, Hamilton, Ontario
  - St. Peter's Chedoke, Hamilton, Ontario
  - Wentworth Lodge, Hamilton, Ontario
  - Blackadar Continuing Care, Hamilton, Ontario
  - St. Joseph's Villa, Hamilton, Ontario

REFERENCES:
- [Derived] Wang B, Hylwka T, Smieja M, Surrette M, Bowdish DME, Loeb M. Probiotics to Prevent Respiratory Infections in Nursing Homes: A Pilot Randomized Controlled Trial. J Am Geriatr Soc. 2018 Jul;66(7):1346-1352. doi: 10.1111/jgs.15396. Epub 2018 May 9. PMID 29741754
- See also: McMaster University, Faculty of Health Sciences, Dr. Mark Loeb — http://mcmaster.ca